CLINICAL TRIAL: NCT05427344
Title: Effectiveness of Cancer Patients' Aquatic Exercise Program for Cancer-related Fatigue, Cancer-related Neuropathy, Activity and Participation, Quality of Life and Return to Work: A Randomized Controlled Trial
Brief Title: Effectiveness of Aquatic Exercise on Fatigue, Neuropathy and Quality of Life Among Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped because we were unable to recruit participants as planned. Therefore, it was decided to halt the study and participant recruitment.
Sponsor: Tel Aviv University (Other)
Collaborators: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Navah Ratzon, Head School of Health Professions Sackler Faculty of Medicine, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Michal Nissim 2
Record Dates: First submitted 2021-10-07; First posted 2022-06-22 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Colon Cancer; Breast Cancer
MeSH Terms: conditions — Colonic Neoplasms; Breast Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water exercise group (Experimental): Water exercise group where the Ai Chi technique was selected as the exercise method of choice. The activity will take place in a hydrotherapy pool approved by the Ministry of Health and will be led by a hydrotherapist who has been trained in Ai Chi
  Interventions: Other: Water exercise group
- Land exercise group (Experimental): Land exercise group who will perform the same Ai Chi movements on land in order to standardize the groups. The activity will take place in a hall and will be led by a physiotherapist who has been trained to teach Ai Chi on land
  Interventions: Other: Land exercise group
- Control group (Experimental): Control group who will not perform additional physical activity or receive any extra treatments
  Interventions: Other: Control group

INTERVENTIONS:
Other: Water exercise group — Water exercise group where the Ai Chi technique was selected as the exercise method of choice. The activity will take place in a hydrotherapy pool approved by the Ministry of Health and will be led by a hydrotherapist who has been trained in Ai Chi.
  Arms: Water exercise group
Other: Land exercise group — Land exercise group who will perform the same Ai Chi movements on land in order to standardize the groups. The activity will take place in a hall and will be led by a physiotherapist who has been trained to teach Ai Chi on land.
  Arms: Land exercise group
Other: Control group — Control group who will not perform additional physical activity or receive any extra treatments.
  Arms: Control group

SUMMARY:
The majority of cancer patients experience exhaustion, fatigue, and neuropathy that impact their participation in daily activities and reduce their quality of life. In addition, they may affect the ability to function at work and delay a return to employment. Studies have demonstrated that physical activity has a positive effect and consequently, patients being treated for cancer are advised to avoid inactivity. Various studies have described Tai Chi practice as beneficial in reducing exhaustion and fatigue to some extent, and have suggested that it may improve the quality of life of cancer patients. The environment in which physical activity takes place is also important. The properties of water and their effect on the submerged human body may be particularly beneficial for cancer patients. A previous study among breast cancer patients reported that exercise in deep water significantly reduced exhaustion and fatigue compared to patients who received only regular treatment. The practice of Tai Chi in water is termed Ai Chi.

The objectives of the present study are to examine the effects of an Ai Chi program as compared to an intervention group undergoing identical physical exercise on land, and a third group with no additional exercise in cancer patients on:(A)time to return to work, work hours, perception of work-related difficulties, and work absenteeism;(B)activity and participation in the daily life and quality of life; and(C)exhaustion, fatigue, and neuropathy.

This is a randomized clinical trial. 150 cancer patients aged 18-65 years will be recruited. Subjects who meet the recruitment criteria will be randomly divided into one of three groups:(a)Water exercise (Ai Chi);(b)Identical land exercise; and(c)Control-who will not perform additional physical activity or receive any extra treatments. The exercise program will be scheduled for 30 minutes twice a week for 8 weeks. Research tools include:(1)WHODAS 2.0;(2)EORTC QLQ-C30; (3)Piper Fatigue Scale;(4) Employment Barriers Questionnaire;(5) Neuropathy Questionnaire (EORTCOLO QLQ-CIPN20);and(6)Date of return to work and duration of working hours - self-report by the study participants.

Data will be collected before the intervention, after 8 weeks of intervention, and then at 3, 12, and 24 months from the end of the intervention. The investigators will perform a series of mixed variance analyzes to identify relationships and associations between groups and with time within a group (independent variables).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer (stage 3 colon cancer patients and breast cancer patients with lymph node involvement). recruitment of colorectal cancer patients and breast cancer patients for the study will be within 3 months of cessation of chemotherapy treatment.
* a score above 26 on the cognitive MOCA test.

Exclusion Criteria:

* Volunteers with orthopedic disabilities / injuries that in the opinion of the attending physician prevent their participation in physical exercise
* Volunteers engaged in other physical activity on a regular basis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-11-23 (Estimated); Study Completion 2024-11-23 (Estimated)

PRIMARY OUTCOMES:
Changes in degree of activity and participation before the start of the intervention (at baseline) and 8 weeks of intervention | Data will be collected before the start of the intervention (at baseline) and 8 weeks of intervention
  WHODAS 2.0 is a self-report questionnaire that captures the level of functioning in six domains of life: Cognition - understanding and communicating, Mobility - moving and getting around, Self-care - attending to one's hygiene, dressing, eating and staying alone, Getting along - interacting with other people, Life activities - domestic responsibilities, leisure, work and school, Participation - joining in community activities, participating in society.
  The average scores are comparable to the WHODAS 5-point scale, which allows the clinician to think of the individual's disability in terms of none (0-0.49), mild (0.5-1.49), moderate (1.5-2.49), severe (2.5-3.49), or extreme (3.5-4). The average domain score is calculated by dividing the raw domain score by the number of items in the domain. The average general disability score is calculated by dividing the raw overall score by number of items in the measure (36). The scoring method is used for each of the 6 domains
Changes in degree of activity and participation before the start of the intervention (at baseline) and 3 months from the end of the intervention. | Data will be collected before the start of the intervention (at baseline) and 3 months from the end of the intervention
  WHODAS 2.0 is a self-report questionnaire that captures the level of functioning in six domains of life: Cognition - understanding and communicating, Mobility - moving and getting around, Self-care - attending to one's hygiene, dressing, eating and staying alone, Getting along - interacting with other people, Life activities - domestic responsibilities, leisure, work and school, Participation - joining in community activities, participating in society.
  The average scores are comparable to the WHODAS 5-point scale, which allows the clinician to think of the individual's disability in terms of none (0-0.49), mild (0.5-1.49), moderate (1.5-2.49), severe (2.5-3.49), or extreme (3.5-4). The average domain score is calculated by dividing the raw domain score by the number of items in the domain. The average general disability score is calculated by dividing the raw overall score by number of items in the measure (36). The scoring method is used for each of the 6 domains
Changes in degree of activity and participation, before the start of the intervention (at baseline), and 12 months from the end of the intervention. | Data will be collected before the start of the intervention (at baseline), and 12, months from the end of the intervention.
  WHODAS 2.0 is a self-report questionnaire that captures the level of functioning in six domains of life: Cognition - understanding and communicating, Mobility - moving and getting around, Self-care - attending to one's hygiene, dressing, eating and staying alone, Getting along - interacting with other people, Life activities - domestic responsibilities, leisure, work and school, Participation - joining in community activities, participating in society.
  The average scores are comparable to the WHODAS 5-point scale, which allows the clinician to think of the individual's disability in terms of none (0-0.49), mild (0.5-1.49), moderate (1.5-2.49), severe (2.5-3.49), or extreme (3.5-4). The average domain score is calculated by dividing the raw domain score by the number of items in the domain. The average general disability score is calculated by dividing the raw overall score by number of items in the measure (36). The scoring method is used for each of the 6 domains
Changes in degree of activity and participation before the start of the intervention (at baseline) and 24 months from the end of the intervention. | Data will be collected before the start of the intervention (at baseline) and 24 months from the end of the intervention.
  WHODAS 2.0 is a self-report questionnaire that captures the level of functioning in six domains of life: Cognition - understanding and communicating, Mobility - moving and getting around, Self-care - attending to one's hygiene, dressing, eating and staying alone, Getting along - interacting with other people, Life activities - domestic responsibilities, leisure, work and school, Participation - joining in community activities, participating in society.
  The average scores are comparable to the WHODAS 5-point scale, which allows the clinician to think of the individual's disability in terms of none (0-0.49), mild (0.5-1.49), moderate (1.5-2.49), severe (2.5-3.49), or extreme (3.5-4). The average domain score is calculated by dividing the raw domain score by the number of items in the domain. The average general disability score is calculated by dividing the raw overall score by number of items in the measure (36). The scoring method is used for each of the 6 domains
Changes in Quality of life before the start of the intervention (at baseline) and 8 weeks of intervention | Data will be collected before the start of the intervention (at baseline) and 8 weeks of intervention
  The EORTC QLQ-C30 has 30 items arranged into nine scales (dimensions) and six single items. The scales are divided into five function scales (physical, role, cognitive, emotional and social functions); three symptom scales (fatigue, pain, nausea or vomiting) and one global health-status/quality of life dimension. The six single items address specific symptoms: dyspnoea, appetite loss, insomnia, constipation, diarrhoea and a question addressing the financial impact of the disease. Each item has four response alternatives: 1) "not at all", 2) "a little" 3) "quite a bit" 4) "very much" except for the global health-status/quality of life scale, which has response options ranging from 1) "very poor" to 7) "excellent".
Changes in Quality of life before the start of the intervention (at baseline) and 3 months from the end of the intervention | Data will be collected before the start of the intervention (at baseline) and 3 months from the end of the intervention
  The EORTC QLQ-C30 has 30 items arranged into nine scales (dimensions) and six single items. The scales are divided into five function scales (physical, role, cognitive, emotional and social functions); three symptom scales (fatigue, pain, nausea or vomiting) and one global health-status/quality of life dimension. The six single items address specific symptoms: dyspnoea, appetite loss, insomnia, constipation, diarrhoea and a question addressing the financial impact of the disease. Each item has four response alternatives: 1) "not at all", 2) "a little" 3) "quite a bit" 4) "very much" except for the global health-status/quality of life scale, which has response options ranging from 1) "very poor" to 7) "excellent".
Changes in Quality of life before the start of the intervention (at baseline) and 12 months from the end of the intervention | Data will be collected before the start of the intervention (at baseline), and 12 months from the end of the intervention.
  The EORTC QLQ-C30 has 30 items arranged into nine scales (dimensions) and six single items. The scales are divided into five function scales (physical, role, cognitive, emotional and social functions); three symptom scales (fatigue, pain, nausea or vomiting) and one global health-status/quality of life dimension. The six single items address specific symptoms: dyspnoea, appetite loss, insomnia, constipation, diarrhoea and a question addressing the financial impact of the disease. Each item has four response alternatives: 1) "not at all", 2) "a little" 3) "quite a bit" 4) "very much" except for the global health-status/quality of life scale, which has response options ranging from 1) "very poor" to 7) "excellent".
Changes in Quality of life before the start of the intervention (at baseline) and 24 months from the end of the intervention | Data will be collected before the start of the intervention (at baseline), and 24 months from the end of the intervention.
  The EORTC QLQ-C30 has 30 items arranged into nine scales (dimensions) and six single items. The scales are divided into five function scales (physical, role, cognitive, emotional and social functions); three symptom scales (fatigue, pain, nausea or vomiting) and one global health-status/quality of life dimension. The six single items address specific symptoms: dyspnoea, appetite loss, insomnia, constipation, diarrhoea and a question addressing the financial impact of the disease. Each item has four response alternatives: 1) "not at all", 2) "a little" 3) "quite a bit" 4) "very much" except for the global health-status/quality of life scale, which has response options ranging from 1) "very poor" to 7) "excellent".
Changes in Exhaustion and fatigue before the start of the intervention (at baseline) and 8 weeks of intervention | Data will be collected before the start of the intervention (at baseline) and 8 weeks of intervention
  Piper Fatigue Scale - to assess the levels of exhaustion and fatigue. It consists of 22 numerical items to assess fatigue at the time of the questionnaire. The items are scored on a 0-10 Likert scale and measure the four dimensions of behavioral/severity (six items), affective meaning (five items), sensory (five items), and cognitive/mood (six items). To calculate the subscale score, the scores of the items on the specific subscales are summed and divided by the number of items in the subscale. All item scores are summed and divided by 22 to calculate the total fatigue score, which has a range from 0 to 10, with a high score indicating a high fatigue level.
Changes in Exhaustion and fatigue before the start of the intervention (at baseline) and 3 months from the end of the intervention. | Data will be collected before the start of the intervention (at baseline) and 3 months from the end of the intervention
  Piper Fatigue Scale - to assess the levels of exhaustion and fatigue. It consists of 22 numerical items to assess fatigue at the time of the questionnaire. The items are scored on a 0-10 Likert scale and measure the four dimensions of behavioral/severity (six items), affective meaning (five items), sensory (five items), and cognitive/mood (six items). To calculate the subscale score, the scores of the items on the specific subscales are summed and divided by the number of items in the subscale. All item scores are summed and divided by 22 to calculate the total fatigue score, which has a range from 0 to 10, with a high score indicating a high fatigue level.
Changes in Exhaustion and fatigue before the start of the intervention (at baseline) and 12 months from the end of the intervention. | Data will be collected before the start of the intervention (at baseline) and 12 months from the end of the intervention
  Piper Fatigue Scale - to assess the levels of exhaustion and fatigue. It consists of 22 numerical items to assess fatigue at the time of the questionnaire. The items are scored on a 0-10 Likert scale and measure the four dimensions of behavioral/severity (six items), affective meaning (five items), sensory (five items), and cognitive/mood (six items). To calculate the subscale score, the scores of the items on the specific subscales are summed and divided by the number of items in the subscale. All item scores are summed and divided by 22 to calculate the total fatigue score, which has a range from 0 to 10, with a high score indicating a high fatigue level.
Changes in Exhaustion and fatigue before the start of the intervention (at baseline) and 24 months from the end of the intervention. | Data will be collected before the start of the intervention (at baseline) and 24 months from the end of the intervention
  Piper Fatigue Scale - to assess the levels of exhaustion and fatigue. It consists of 22 numerical items to assess fatigue at the time of the questionnaire. The items are scored on a 0-10 Likert scale and measure the four dimensions of behavioral/severity (six items), affective meaning (five items), sensory (five items), and cognitive/mood (six items). To calculate the subscale score, the scores of the items on the specific subscales are summed and divided by the number of items in the subscale. All item scores are summed and divided by 22 to calculate the total fatigue score, which has a range from 0 to 10, with a high score indicating a high fatigue level.
Changes in Employment before the start of the intervention (at baseline) and 8 weeks of intervention | Data will be collected before the start of the intervention (at baseline) and 8 weeks of intervention
  Employment Barriers Questionnaire. It consists of 77 numerical items to assess workers barriers at the time of the questionnaire. The items are scored on a 0-4 Likert scale and measure the two dimensions of environmental and occupational barriers.
Changes in Employment before the start of the intervention (at baseline) and 3 months from the end of the intervention. | Data will be collected before the start of the intervention (at baseline) and 3 months from the end of the intervention
  Employment Barriers Questionnaire. It consists of 77 numerical items to assess workers barriers at the time of the questionnaire. The items are scored on a 0-4 Likert scale and measure the two dimensions of environmental and occupational barriers.
Changes in Employment before the start of the intervention (at baseline) and 12 months from the end of the intervention. | Data will be collected before the start of the intervention (at baseline) and 12 months from the end of the intervention
  Employment Barriers Questionnaire. It consists of 77 numerical items to assess workers barriers at the time of the questionnaire. The items are scored on a 0-4 Likert scale and measure the two dimensions of environmental and occupational barriers.
Changes in Employment before the start of the intervention (at baseline) and 24 months from the end of the intervention. | Data will be collected before the start of the intervention (at baseline) and 24 months from the end of the intervention
  Employment Barriers Questionnaire. It consists of 77 numerical items to assess workers barriers at the time of the questionnaire. The items are scored on a 0-4 Likert scale and measure the two dimensions of environmental and occupational barriers.
Changes in Neuropathy before the start of the intervention (at baseline) and 8 weeks of intervention | Data will be collected before the start of the intervention (at baseline) and 8 weeks of intervention
  Neuropathy Questionnaire (EORTCOLO QLQ-CIPN20). This is a 20-item patient self-report CIPN-specific questionnaire that includes three subscales assessing sensory, motor, and autonomic symptoms with each item measured on a 1-4 Likert scale (1 being "not at all" and 4 being "very much"). Items in the sensory subscale inquire about tingling, numbness, and shooting/burning pain separately for (1) fingers and hands as well as (2) toes and feet.
Changes in Neuropathy before the start of the intervention (at baseline) and 3 months from the end of the intervention. | Data will be collected before the start of the intervention (at baseline) and 3 months from the end of the intervention
  Neuropathy Questionnaire (EORTCOLO QLQ-CIPN20). This is a 20-item patient self-report CIPN-specific questionnaire that includes three subscales assessing sensory, motor, and autonomic symptoms with each item measured on a 1-4 Likert scale (1 being "not at all" and 4 being "very much"). Items in the sensory subscale inquire about tingling, numbness, and shooting/burning pain separately for (1) fingers and hands as well as (2) toes and feet.
Changes in Neuropathy before the start of the intervention (at baseline) and 12 months from the end of the intervention. | Data will be collected before the start of the intervention (at baseline) and 12 months from the end of the intervention
  Neuropathy Questionnaire (EORTCOLO QLQ-CIPN20). This is a 20-item patient self-report CIPN-specific questionnaire that includes three subscales assessing sensory, motor, and autonomic symptoms with each item measured on a 1-4 Likert scale (1 being "not at all" and 4 being "very much"). Items in the sensory subscale inquire about tingling, numbness, and shooting/burning pain separately for (1) fingers and hands as well as (2) toes and feet.
Changes in Neuropathy before the start of the intervention (at baseline) and 24 months from the end of the intervention. | Data will be collected before the start of the intervention (at baseline) and 24 months from the end of the intervention
  Neuropathy Questionnaire (EORTCOLO QLQ-CIPN20). This is a 20-item patient self-report CIPN-specific questionnaire that includes three subscales assessing sensory, motor, and autonomic symptoms with each item measured on a 1-4 Likert scale (1 being "not at all" and 4 being "very much"). Items in the sensory subscale inquire about tingling, numbness, and shooting/burning pain separately for (1) fingers and hands as well as (2) toes and feet.
Changes in duration of working hours before the start of the intervention (at baseline) and 8 weeks of intervention | Data will be collected before the start of the intervention (at baseline) and 8 weeks of intervention
  Duration of working hours - self-report by the study participants
Changes in duration of working hours before the start of the intervention (at baseline) and 3 months from the end of the intervention. | Chang in Employment before the start of the intervention (at baseline) and 3 months from the end of the intervention.
  Duration of working hours - self-report by the study participants
Changes in duration of working hours before the start of the intervention (at baseline) and 12 months from the end of the intervention. | Chang in Employment before the start of the intervention (at baseline) and 12 months from the end of the intervention.
  Duration of working hours - self-report by the study participants
Changes in duration of working hours before the start of the intervention (at baseline) and 24 months from the end of the intervention. | Chang in Employment before the start of the intervention (at baseline) and 24 months from the end of the intervention.
  Duration of working hours - self-report by the study participants

CONTACTS AND LOCATIONS:
Overall Officials: Navah Z Ratzon, Prof, Principal Investigator — Tel Aviv University
Locations (1):
- Hadassa Hospital, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nissim M, Rottenberg Y, Karniel N, Ratzon NZ. Effects of aquatic exercise program versus on-land exercise program on cancer-related fatigue, neuropathy, activity and participation, quality of life, and return to work for cancer patients: study protocol for a randomized controlled trial. BMC Complement Med Ther. 2024 Feb 2;24(1):74. doi: 10.1186/s12906-024-04367-8. PMID 38308248